CLINICAL TRIAL: NCT02290613
Title: Early Treatment of Borderline Pulmonary Arterial Hypertension Associated With Systemic Sclerosis (SSc-APAH) A Randomized, Controlled, Double-blind, Parallel Group, Proof-of-concept Trial EDITA
Brief Title: Early Treatment of Borderline Pulmonary Arterial Hypertension Associated With Systemic Sclerosis (SSc-APAH)
Acronym: EDITA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-05ED
Record Dates: First submitted 2014-10-31; First posted 2014-11-14 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Systemic Sclerosis; Pulmonary Hypertension
Keywords: pulmonary hypertension; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambrisentan Verum (Experimental): Study medication will be ambrisentan 10 mg (starting with 5 mg in the beginning of the study and then up-titrated to 10 mg/day).
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Titration:
  As common practice of the clinic, the patient will adapt the dose from 5 mg to 10 mg after 1 to 4 weeks according to tolerability and after consultation (by phone or personally) with one of the investigators.
  Additionally, at each study visit the investigator needs to decide, based on the patient's well-being, patients´ assessment, safety parameters, and tolerance of ambrisentan, if the study medication should be modified. The respective decision (increase, maintain or decrease dose) must be documented.
  Maximum dose allowed: not to exceed 10 mg/day.
  Administration:
  Ambrisentan and placebo will be administered orally with or without food intake.
  Other Names: Volibris; ATC code: C02KX02
  Arms: Ambrisentan Verum
Drug: Placebo — Placebo tablet (one to two tablets corresponding to one to two verum tablets)
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
Trial Design Patients with borderline PAH indicated by borderline mPAP values will be included in this single centre study. This clinical investigation is performed as a Proof-of-Concept (PoC) investigator initiated trial (IIT) using a prospective, randomized, double-blind, parallel group, placebo-controlled, phase IIA clinical study design. On their first visit their medical history will be obtained and physical examination will be conducted. Moreover, an electrocardiogram (ECG), laboratory testing (NT-proBNP, uric acid and other laboratory tests), echocardiography at rest and right heart catheterization will be carried out. If patients have been identified within the last 6 months before screening investigations by right heart catheterization, the measurements are considered valid as baseline investigations and will not be repeated. If patients fulfill the inclusion criteria and still suffer from borderline mPAP values they will be invited to join the study. The clinical investigations will begin within 28 days. The prospective study will comprise a 6 months study period (180 ±2 weeks) plus the screening phase up to 28 days and a follow-up phase of 30 ±7 days.

DETAILED DESCRIPTION:
Treatment naïve patients with SSc-APAH will be included in the investigator initiated trial (IIT) to assess efficacy and safety of ambrisentan. As patients life-expectancy after diagnosis of untreated patients is only one year we put forward a screening to identify borderline PAH patients and treat them before PH manifests. Therapy with ambrisentan reached a significant improvement in SSc-IPAH patients (Galiè et al. 2008). In PAH mPAP improved about 15% due to ambrisentan (Klinger et al. 2011).

Thus, especially patients with SSc-APAH have a high need for an early diagnosis and therapy. It is important to determine factors predictive of incident SSc-APAH and PH as well as the event rate of PAH and PH occurrence. Early identification and intervention with specific modern therapies as with ambrisentan may improve hemodynamic, symptoms, exercise capacity, quality of life and outcomes in this patient population, in particular in SSc-patients of borderline-PAH. It is considered reasonable that the development of manifest APAH might be preventable in this defined population with SSc and early pulmonary vascular changes. A reliable trial testing this latter hypothesis cannot be performed without critical evidence which defines the response to medical PAH-targeted therapy in borderline-PAH and the associated disease progression of manifest PAH.

Due to the positive results in the treatment of patients with SSc-APAH, the initiation of this proof-of-concept study is justified.

Previously identified patients with borderline PAH indicated by borderline mPAP values will be included in this single centre randomized, controlled, double-blind, parallel group, proof-of-concept (PoC) phase IIa IIT. If assessments necessary for screening have already been made under the screening for PH in Systemic sclerosis trial (non-drug trial, Ethics committee of Heidelberg # S360/2009), these examinations may be used for screening for this trial, as long as they have been performed within the given time frame of the screening period.

On their first visit the patients' medical history will be obtained and physical examination will be conducted. Moreover, an electrocardiogram (ECG), laboratory testing (NT-proBNP, uric acid and other laboratory tests), echocardiography at rest and during exercise and right heart catheterization will be carried out. If patients fulfill the inclusion criteria and still suffer from borderline mPAP values they will be invited to join the study. Patients will be asked to sign the informed consent form (ICF) before the initial screening will be conducted. Randomization will be performed after a maximum of 28 days and medication or placebo will be provided. If patients have been identified within the last 6 months before baseline by right heart catheterization, the measurements are considered valid for the baseline visit to spare patients a repetition of this invasive procedure. Non-invasive measurements that are out of the time-frame have to be repeated for the study. An 1:1 oral ambrisentan: oral Placebo randomization will be performed.

Patients will be randomized into either:

* A treatment arm with ambrisentan treatment (19 patients)
* A placebo arm (19 patients will receive placebo). Safety and tolerability will be controlled at each study visit until the end of study (day 180 ± 2 weeks). If necessary, the dose will be adapted. As to common practice of the clinic, the patient will adapt the dose according to tolerability and after consultation (by phone or personally) with one of the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. mPAP 21-24 mmHg, TPG > 11mmHg, PAWP <15 mmHg and/or
2. Exercise induced elevated mPAP-values >30 mmHg, PAWP <18 mmHg; TPG >15 mmHg, as defined in Saggar et al. (2012) without left heart or severe lung disease or systemic arterial hypertension
3. Adult patients having completed his/her 18th birthday
4. Patients with definite diagnosis of Systemic Sclerosis using the scleroderma criteria of the American Rheumatism Association
5. SSc-disease duration >3 years
6. Able to understand and willing to sign the Informed Consent Form
7. Negative pregnancy test at the start of the trial and appropriate contraception throughout the study for women with child-bearing potential.

Exclusion Criteria:

1. Any connective tissue diseases (CTD) other than SSc
2. Pulmonary hypertension (PH) confirmed by right heart catheter (RHC) before enrolment, i.e. mPAP ≥25 mmHg at rest
3. Patients presenting normal mPAP values, that is mPAP<21 mmHg at rest, ≤30 mmHg during exercise, PAWP >=15 mmHg at rest or <=18 mmHg during exercise
4. Ongoing or a history of >2 weeks of continued use of therapies that are considered definitive PH treatment: endothelin receptor antagonists (ERA; e.g. bosentan, ambrisentan), phosphodiesterase type 5 inhibitors (PDE5; e.g. sildenafil, tadalafil, vardenafil), prostanoids (e.g. epoprostenol, treprostinil, iloprost, beraprost) and soluble guanylate cyclase stimulator (e.g. Riociguat). Intermittent use of PDE5 inhibitors for male erectile dysfunction is permitted.
5. Except for diuretics and corticosteroids medical treatment should not be expected to change 4 weeks prior inclusion into the study and during the entire 12-week study period.
6. Known intolerance to ambrisentan or one of its excipients
7. Clinically significant anemia (hemoglobin concentration of less than 75% of the lower limit of normal, LLN)
8. Forced vital capacity (FVC) <60%, forced expiratory volume in first second (FEV1) <65%
9. Severe interstitial lung disease, idiopathic pulmonary fibrosis
10. Renal insufficiency (glomerular filtration rate [GFR] <60 mL/min/1.73m2 for at least 3 months)
11. Baseline values of hepatic aminotransferases (ALT and/or AST) >3 x upper limit of normal (ULN)
12. Systolic blood pressure <85 mmHg;
13. evidence of inadequately treated blood pressure >160/90 mmHg and/or blood pressure during exercise >220/120 mmHg
14. Patients referred with clinically significant overt heart failure
15. Clinically significant fluid retention
16. Previous evidence or diagnosis of clinically relevant left heart disease, i.e. at least one of the following: Previous echocardiography with estimated left ventricular (LV) ejection fraction <50%, previous history of cardiogenic pulmonary edema, increased size of left atrium (>50 mm)
17. Known significant diastolic dysfunction associated with clinical heart failure
18. Known coronary disease or significant valvular heart disease
19. Known congenital heart defects such as single ventricle, transposition, Eisenmenger
20. Known hypertrophic cardiomyopathy or left ventricular hypertrophy (interventricular septum thickness (IVS) or posterior wall thickness (PWD) >1.2 cm)
21. Participation in any clinical drug trial within 4 weeks prior to screening of this study and/or who is scheduled to receive another investigational medicinal product (IMP) during the course of this study
22. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekkehard Grünig, MD, Principal Investigator — Thoraxclinic at the University of Heidelberg
Locations (1):
- Thoraxclinic at the University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Galie N, Olschewski H, Oudiz RJ, Torres F, Frost A, Ghofrani HA, Badesch DB, McGoon MD, McLaughlin VV, Roecker EB, Gerber MJ, Dufton C, Wiens BL, Rubin LJ; Ambrisentan in Pulmonary Arterial Hypertension, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Efficacy Studies (ARIES) Group. Ambrisentan for the treatment of pulmonary arterial hypertension: results of the ambrisentan in pulmonary arterial hypertension, randomized, double-blind, placebo-controlled, multicenter, efficacy (ARIES) study 1 and 2. Circulation. 2008 Jun 10;117(23):3010-9. doi: 10.1161/CIRCULATIONAHA.107.742510. Epub 2008 May 27. PMID 18506008
- [Background] Klinger JR, Oudiz RJ, Spence R, Despain D, Dufton C. Long-term pulmonary hemodynamic effects of ambrisentan in pulmonary arterial hypertension. Am J Cardiol. 2011 Jul 15;108(2):302-7. doi: 10.1016/j.amjcard.2011.03.037. Epub 2011 May 3. PMID 21545989
- [Derived] Pan Z, Marra AM, Benjamin N, Eichstaedt CA, Blank N, Bossone E, Cittadini A, Coghlan G, Denton CP, Distler O, Egenlauf B, Fischer C, Harutyunova S, Xanthouli P, Lorenz HM, Grunig E. Early treatment with ambrisentan of mildly elevated mean pulmonary arterial pressure associated with systemic sclerosis: a randomized, controlled, double-blind, parallel group study (EDITA study). Arthritis Res Ther. 2019 Oct 26;21(1):217. doi: 10.1186/s13075-019-1981-0. PMID 31655622

RESULTS

PARTICIPANT FLOW:
Groups:
- Ambrisentan Verum: Study medication will be ambrisentan 10 mg (starting with 5 mg in the beginning of the study and then up-titrated to 10 mg/die).
  Ambrisentan: Titration:
  As common practice of the clinic, the patient will adapt the dose from 5 mg to 10 mg after 1 to 4 weeks according to tolerability and after consultation (by phone or personally) with one of the investigators.
  Additionally, at each study visit the investigator needs to decide, based on the patient's well-being, patients´ assessment, safety parameters, and tolerance of ambrisentan, if the study medication should be modified. The respective decision (increase, maintain or decrease dose) must be documented.
  Maximum dose allowed: not to exceed 10 mg/die.
  Administration:
  Ambrisentan and placebo will be administered orally with or without food intake.
Period: Overall Study
Arm/Group | Ambrisentan Verum | Placebo
Started | 19 | 19
Completed | 17 | 15
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan Verum | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.8) | 54.9 (11.2) | 56.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of SSc [Count of Participants; unit: Participants]
  dcSSc | 4 | 11 | 15
  lcSSc | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Pulmonary Arterial Pressure Change From Baseline
Description: Determine whether mean pulmonary arterial pressure of SSc patients with borderline - PAH (mPAP 21 24 mmHg, TPG >11 mmHg) can be reduced by 3 mm Hg (absolute change baseline vs. 6 months; equals 15%) following treatment with ambrisentan 10 mg/die (initiated with 5 mg/die and elevated up to 10 mg/die) over 6 months (primary endpoint) compared to baseline and placebo.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
mmHg | -1.0 (6.4) | -0.73 (3.6)

2. Secondary Outcome: Mean Pulmonary Arterial Pressure During Exercise Change From Baseline
Description: Determine whether exercise induced elevated mean pulmonary arterial pressure-values (>30 mmHg without left heart or severe lung disease or systemic arterial hypertension) can be reduced by ambrisentan 10 mg/die over 6 months.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 15 | 13
mmHg | -0.73 (6.23) | 1.08 (7.39)

3. Secondary Outcome: 6-Minute-walking Test
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
meters | 21.53 (34.6) | -16.53 (77.32)

4. Secondary Outcome: Borg Dyspnea Index
Description: measured directly after 6 minute walking distance; The Borg dyspnea index is an standardized scale which reports the subjective feeling of exertion from 0 (no dyspnea) to 10 (maximal feeling of dyspnea).
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
units on a scale | 0.62 (1.7) | 0.08 (1.54)

5. Secondary Outcome: Quality of Life (SF-36) Questionnaire
Description: SF-36 Questionnaire; physical Summation score; All scores and subscores of the SF-36 questionnaire range from 0 (low quality of life) to 100 (high quality of life). The physical Summation score is a compound score including the physical dimensions of the SF-36.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
units on a scale | -6.71 (12.17) | 0.87 (16.01)

6. Secondary Outcome: Lung Function
Description: DLCo (diffusing capacity or transfer factor of the lung for carbon monoxide (CO))
Time Frame: baseline,6 months
Measure: Mean (Standard Deviation); unit: % of target value
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 13
% of target value | 1.19 (1.81) | -0.44 (1.84)

7. Secondary Outcome: Lung Function
Description: DLCo (diffusing capacity or transfer factor of the lung for carbon monoxide (CO))
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmol/min/kPa
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
mmol/min/kPa | -0.32 (1.44) | -0.45 (1.70)

8. Secondary Outcome: Lung Function
Description: FVC (forced vital capacity)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: % of target
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
% of target | -3.31 (5.56) | -1.04 (5.60)

9. Secondary Outcome: Lung Function
Description: FEV1 (forced expiratory volume in one second)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 16 | 15
Litres | -0.11 (0.21) | -0.06 (0.20)

10. Secondary Outcome: Lung Function
Description: TLC (total lung capacity)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 16 | 15
Litres | -0.06 (0.37) | -0.03 (0.36)

11. Secondary Outcome: Lung Function
Description: residual volume
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 16 | 15
Litres | -0.03 (0.33) | 0.05 (0.37)

12. Secondary Outcome: Echocardiography
Description: RA-area (right atrial area)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
cm^2 | 1.65 (2.67) | -0.47 (4.07)

13. Secondary Outcome: Echocardiography
Description: RV-area (right ventricular area)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
cm^2 | -0.15 (3.46) | -0.8 (3.05)

14. Secondary Outcome: Echocardiography
Description: TAPSE (tricuspid annular plane systolic excursion)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
cm | 0.12 (0.41) | -0.19 (0.54)

15. Secondary Outcome: Echocardiography
Description: sPAP (systolic pulmonary arterial pressure)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
mmHg | -0.82 (4.46) | -0.93 (6.08)

16. Secondary Outcome: WHO-functional Class
Description: The World Health Organization functional class includes four categories with
  1. Patients with Pulmonary Hypertension but without any resulting limitation of physical activity.
  2. Patients with Pulmonary Hypertension resulting in slight limitation of physical activity.
  3. Patients with Pulmonary Hypertension resulting in marked limitation of physical activity.
  4. Patients with pulmonary hypertension with inability to carry out any physical activity without symptoms.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
Participants
  FC II | 17 | 13
  FC III | 0 | 2

17. Secondary Outcome: Hemodynamics
Description: right atrial pressure
Time Frame: change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
mmHg | 0.82 (4.11) | -0.2 (2.76)

18. Secondary Outcome: Hemodynamics
Description: pulmonary vascular resistance
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: Wood Units
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
Wood Units | -0.59 (0.79) | 0.02 (0.76)

19. Secondary Outcome: Hemodynamics
Description: cardiac output (CO)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
L/min | 0.58 (1.17) | -0.26 (1.11)

20. Secondary Outcome: Hemodynamics
Description: cardiac index (CI)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 16 | 15
L/min/m^2 | 0.36 (0.66) | -0.31 (0.71)

21. Secondary Outcome: Hemodynamics
Description: PAWP (pulmonary arterial wedge pressure)
Time Frame: baseline , 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 17 | 15
mmHg | 1.24 (5.31) | 0.13 (3.20)

22. Secondary Outcome: Hemodynamics
Description: venous oxygen saturation (SvO2)
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: % saturation
Arm/Group | Ambrisentan Verum | Placebo
Number analyzed (Participants) | 12 | 13
% saturation | -2.79 (7.56) | -3.48 (12.26)

ADVERSE EVENTS:
Time Frame: adverse Events were collected throughout the study from baseline to the 6 month-assessment and 30 days follow-up.
Arm/Group | Ambrisentan Verum | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/19 | 5/19
Other Adverse Events (participants affected / at risk) | 17/19 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan Verum (N=19) | Placebo (N=19)
Lower jaw fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphangitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Raynaud (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan Verum (N=19) | Placebo (N=19)
Headache (Nervous system disorders) | 6 (6) | 6 (6)
Edema (Cardiac disorders) | 8 (8) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 4 (4) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3)
arterial hypotension (Cardiac disorders) | 2 (2) | 2 (2)
Epistaxis (Vascular disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT02290613/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT02290613/SAP_001.pdf